CLINICAL TRIAL: NCT04822246
Title: Excavation of Root Caries with Air-water Powder Stream Vs Manual Excavation for Atraumatic Restorative Treatment in Older Patients: a Single-blind Randomized Controlled Trial
Brief Title: Root Caries Excavation with Air Water/powder Prophylaxis Device for ART Restorations
Acronym: ART-AIRFLOW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murali Srinivasan, Dr. med. dent., BDS, MDS, MBA, MAS (Other)
Responsible Party: Sponsor-Investigator, Murali Srinivasan, Dr. med. dent., BDS, MDS, MBA, MAS, Prof., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UZH_ABS_2021_4
Record Dates: First submitted 2021-03-16; First posted 2021-03-30 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Dental Caries Extending Into Dentin; Root Caries
Keywords: Root caries; Elders; Atraumatic restorative treatment; Glass-ionomer cement
MeSH Terms: conditions — Root Caries | interventions — Powders

STUDY DESIGN:
Intervention Model Description: Single-blind, RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control: Hand instrumentation for caries excavation (Other): Hand instrumentation for caries excavation
  Interventions: Procedure: Control: Hand instrumentation for caries excavation
- Intervention 1: EMS Airflow device for caries excavation (Experimental): Powder/water jet prophylaxis device (EMS Airflow) for caries excavation
  Interventions: Procedure: Intervention 1: EMS Airflow device for caries excavation
- Intervention 2: Hand excavation + EMS Airflow device for caries excavation (Experimental): Hand excavation and Powder/ jet prophylaxis device (EMS Airflow) for caries excavation
  Interventions: Procedure: Intervention 2: Hand excavation + EMS Airflow device for caries excavation

INTERVENTIONS:
Procedure: Control: Hand instrumentation for caries excavation — An enamel hatchet will be used to create access to the carious lesion and then removal of soft carious tissue will be undertaken with excavators. Excavation will be stopped when some resistance to excavation will be felt and the cavity will be then conditioned with polyacrylic acid for 20 s, washed and dried with cotton pellets. A high-viscosity glass-ionomer cement will be used to restore the cavity. Moisture control will be achieved with the use of cotton wool rolls. A chair-side assistant will hand-mix the glass-ionomer according to manufacturers' instructions and it will be placed in the cavity using the "press-finger" technique whenever the type of cavity allows it. In the case of root restorations, a glove coated with petroleum jelly will be used similarly to the "press-finger" technique to better condense the material into the cavity. Excess material will be removed; the restoration will be coated with petroleum jelly. No local anaesthetic will be used to provide ART treatment.
  Other Names: Hand instrumentation for caries excavation
  Arms: Control: Hand instrumentation for caries excavation
Procedure: Intervention 1: EMS Airflow device for caries excavation — An enamel hatchet will first be used to gain access into the cavity. Then the powder-water prophylaxis device will be used for the removal of soft carious tissue with the sodium bicarbonate powder-water jet. Excavation will be stopped when the colour of the lesion begins to darken and all the soft deposits are evacuated. The excavation will be done intermittently allowing sufficient time to check with hand instrument the surface hardness of the lesion. If the lesion is still soft excavation will be continued until the surface is hard suitable for restoring. The cavity will be then rinsed with copious water spray to evacuate all the powder-water material. The restoration procedure with a glass-ionomer cement will be done following the same procedures as in the control group.
  Other Names: Powder/water jet prophylaxis device (EMS Airflow) for caries excavation
  Arms: Intervention 1: EMS Airflow device for caries excavation
Procedure: Intervention 2: Hand excavation + EMS Airflow device for caries excavation — The participants allocated to this group will have the caries excavated as described for the control group. Then prior to filling the excavated cavity, the procedure of sodium bicarbonate powder-water jet irrigation as described for the intervention group #1 will be performed to condition the prepared excavated cavity. Then the restorative procedure will be completed with the restorative material and procedures as described for the previous groups.
  Other Names: Hand excavation and Powder/ jet prophylaxis device (EMS Airflow) for caries excavation
  Arms: Intervention 2: Hand excavation + EMS Airflow device for caries excavation

SUMMARY:
The main objective of this RCT is to compare the efficacy of a powder/water jet prophylaxis device and conventional hand excavation in excavating root surface caries, with regard to restoration survival/success in older adults.

The secondary outcome of this RCT is to assess the participants' treatment preferences for the received treatment with regard to the procedures involved and in the invasiveness of the procedures carried out during the ART restoration.

ELIGIBILITY:
Inclusion criteria

* Adults ≥65 years
* Dentinal root caries lesions with no painful symptomology
* Can follow instructions for oral hygiene
* Not dependent for care for their ADLs.

Exclusion criteria:

* Symptomatic carious teeth
* Non-carious attrition, erosion or abrasion cavities
* Periodontally compromised teeth with Grade 3 mobility, and active signs of infections.
* Not willing or able to sign informed consent

Post-hoc exclusion:

* Participant withdraws consent
* Medical reasons.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Restoration Success rate | 1 year, year 1
  Restoration success rate (SxR %): For the purpose of this trial, a successful restoration is defined as one that has undergone no changes in its surface / structural integrity, still adhered to the structure and is functional when examined during the scheduled or unscheduled recall visit. The restoration success rate (SxR %) is calculated by the number of successful restorations present at the end of the trial (nsx) divided by the number of restorations placed in the beginning of the trial (N0) multiplied by 100 using the formula: SxR % = (nsx / N0) * 100.
Restoration survival rate | 1 year, year 1
  Restoration survival rate (SvR %): For the purpose of this trial, any restoration, where the surface or structural integrity is compromised, but still adhering to the tooth, is functional and does not warrant a repair or replacement when examined during the scheduled or unscheduled recall visit, is considered survived. The restoration survival rate (SvR %) is calculated by the number of survived restorations present at the end of the trial (nsv) divided by the number of restorations placed in the beginning of the trial (N0) multiplied by 100 using the formula: SvR = (nsv / N0) * 100.

SECONDARY OUTCOMES:
Participants' Treatment preference | Through study completion, an average of 1 year
  Secondary assessment will be to assess the participants' treatment preference. This is done by administering a simple questionnaire which inquires on their treatment preferences.
  After treatment will be completed the dental nurse will question the participant about their treatment preference. The questions will include preferences for restorative treatment with or without the use of anaesthesia, with or without rotary instrumentation, hand instrumentation or with air-water prophylaxis device, compared to their previous dental experience. The response "no difference" will also an option.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic of General, Special care, and Geriatric Dentistry, Center for Dental Medicine, University of Zurich, Zurich, Switzerland